CLINICAL TRIAL: NCT06764238
Title: Chinese Children's Cancer Group-2025 Protocol for Newly Diagnosed for Intermediate/High Risk Childhood B-cell ALL
Brief Title: Newly-diagnosed Intermediate/High Risk Pediatric B-cell ALL Protocol
Acronym: CCCG-I/HR-ALL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024068
Record Dates: First submitted 2024-12-20; First posted 2025-01-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia ALL; Childhood Leukemia, Acute Lymphoblastic; B Cell Acute Lymphoblastic Leukemia (B-ALL)
Keywords: blinatimomab; venetoclax
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — blinatumomab; Methotrexate; venetoclax; Cyclophosphamide; Vincristine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): After PVDL+CAT induction remission phase, patients randomized to Group A will be subjected to consolidation phase with continuous 28 days' blinatumomab followed by 3 cycles of high-dose methotrexate (HDMTX)
  Interventions: Drug: Blinatumomab (Group A)
- Group B (Experimental): After PVDL+CAT induction remission phase, patients randomized to Group B will be subjected to consolidation phase with two 14-day cycles of blinatumomab, alternating with 3 cycles of high-dose methotrexate (HDMTX).
  Interventions: Drug: Blinatumomab (Group B)
- NonRandonmized Group (Experimental): Patients who will not be subjected to blinatomomab randomization, will received PVDL + Venetoclax + mini-hyperCVD as induction phase , subsequently receiving CAT as early intensification.
  Interventions: Drug: Venetoclax (nonRand Group)

INTERVENTIONS:
Drug: Blinatumomab (Group A) — For Group A I/HR-ALL patients after induction remission phase, continuous 28 days' blinatumomab followed by 3 cycles of high-dose methotrexate (HDMTX) will be applied, subsequently followed by interim continuation, late intensification, and maintenance therapy
  Other Names: high-dose methotrexate
  Arms: Group A
Drug: Venetoclax (nonRand Group) — For I/HR patients non eligible for blinatumomab randomization, venetoclax+ mini-hyperCVD will be applied after PVDL induction, subsequently followed by CAT as intensification, interim continuation, late intensification, and maintenance therapy
  Other Names: cyclophosphamide; vincristine; dexamethasone
  Arms: NonRandonmized Group
Drug: Blinatumomab (Group B) — For Group B I/HR-ALL patients after induction remission phase: a two 14-day cycles of blinatumomab, alternating with three cycles of HDMTX will be applied, subsequently followed interim continuation, late intensification, and maintenance therapy
  Other Names: high-dose methotrexate
  Arms: Group B

SUMMARY:
Building upon the results from the CCCG-ALL-2015, CCCG-ALL-2020 multicenter study cohort, concurrent research findings, and the latest clinical trials, the CCCG-ALL-2025 I/HR-B-ALL is thus developed to further improve the event-free survival (EFS), and overall survival (OS), and quality of life (QoL) of children with intermediate- and high- risk B-cell childhood acute lymphoblastic leukaemia (I/HR-B-ALL), while decreasing adverse reactions and transplantation rates. This trial primarily aims to explore:

1. The efficacy of two randomized Blinatumomab application scheme on I/HR-ALL as determined by MRD negatvitiy rate.
2. The efficacy of modified mini-hyperCVD + Venetoclax in I/HR-ALL cannot afford blinatumomab, in contrast to historical control as determined by MRD negatvitiy rate.

DETAILED DESCRIPTION:
The study shown above will lead to the following revisions to the CCCG-ALL2025 I/HR-B-ALL plan, which will be based on the CCCG-ALL2020 plan.

1. After the induction remission phase, all I/HR-B-ALL patients can afford blinatumomab will participate in a blinatumomab+HDMTX randomized controlled trial as consolidation.
2. For patients cannot afford blinatumomab will be treated with venetoclax + modified mini-hyperCVD during the induction phase, then subsequently with CAT as consolidation phase. CAT will removed from induction phase.
3. For patients who received blinatumomab randomization, the CAT+ course was canceled.
4. All patients will continued with 6 cycles of alternated 5-day venetoclax or Dauno-based CCCG-2020 continuous therapy regimen.
5. Adding IgH rearrangement NGS MRD as an evaluation indicator.
6. Adding pharmacotyping study for I/HR B-ALL.
7. Three more bone marrow punctures and IT will be added with the aims to evaluate the CR rate with deepen remission during or after consolidation.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 1 month to younger than 18 years.
2. Diagnosis of acute lymphoblastic leukemia by bone marrow morphology.
3. Diagnosis of B-ALL by immunophenotyping.

Exclusion Criteria:

1. Low-risk ALL
2. sIgM+
3. Acute leukemias of ambiguous lineage diagnosed according to WHO or EGIL criteria.
4. ALL evolved from chronic myeloid leukemia (CML).
5. Down's syndrome, or major congenital or hereditary disease with organ dysfunction
6. Secondary leukemia
7. Known underlying congenital immunodeficiency or metabolic disease
8. Congenital heart disease with cardiac insufficiency.
9. Treated with glucocorticoids for ≥14 days, or ABL kinase inhibitors for > 7 days within one month before enrollment, or any chemotherapy or radiotherapy within 3 months before enrollment (except for emergency radiotherapy to relieve airway compression)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
To investigate if Group B[2*(14-day blinatumomab + HDMTX*2)] can result in noninferior event-free survival (EFS) compared to Group A [28-day blinatumomab + HDMTX*4 | Based on the above analysis in this study the investigators will randomize 1800 patients. The analysis will start1.5 years after the last patient is randomized. The expected study duration is approximately 6.5 years.
  * The randomization is stratified by hospitals and status of flow-cytometry MRD (positive or negative) immediately prior to the blinatumomab-HDMTX treatment.
  * Kaplan-Meier (KM) estimates of each EFS function will be computed along with standard error by the default procedure in R. To test noninferiority the investigators consider a noninferiority margin of 0.04 for 5-year EFS as clinically meaningful.
  * Assume the EFS in the control group (Arm A) to be the same as the provisional I/HR in the CCCG-ALL2020 trial (preliminary data above), with the 1-year and 3-year EFS possibly 0.837 and 0.768 respectively. A simulation study with 10,000 rounds shows that by randomizing 1800 patients and 1.5 years of follow up, the above decision rule of declaring noninferiority has well controlled probabilities of false positive and false negative errors.

SECONDARY OUTCOMES:
Event-free survival (EFS) in the two randomized arms [2*(14-day blinatumomab + HDMTX*2)] and [28-day blinatumomab + HDMTX*4], in contrast to historical regimens. | Up to 5 years for every enrolled case
  EFS functions will be estimated using the Kaplan-Meier estimator of survival functions along with 95% confidence interval at 5 year. Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of EFS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
Cumulative incidence of relapse (CIR) in the two randomized arms [2*(14-day blinatumomab + HDMTX*2)] and [28-day blinatumomab + HDMTX*4], in contrast to historical regimen. | Up to 5 years for every enrolled case
  CIR functions of relapse will be estimated by the Kalbafleisch-Prentice method. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of CIR will be performed by Gray's test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Fine-Gray models.
Overall survival (OS) in the two randomized arms [2*(14-day blinatumomab + HDMTX*2)] and [28-day blinatumomab + HDMTX*4], in contrast to historical regimens. | Up to 5 years for every enrolled case
  OS functions will be estimated using the Kaplan-Meier estimator of survival functions along with 95% confidence interval at 5 year. Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of OS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
EFS in patients who receive 6 alternated venetoclax/Daunorubincin courses of interim continuation therapy. | Up to 5 years for every enrolled case
  EFS functions will be estimated using the Kaplan-Meier estimator of survival functions along with 95% confidence interval at 5 year. Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of EFS will be performed using two-sided log-rank test.Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
CIR in patients who receive 6 alternated venetoclax/Daunorubincin courses of interim continuation therapy. | Up to five years for every enrolled case
  CIR functions of relapse will be estimated by the Kalbafleisch-Prentice method. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of CIR will be performed by Gray's test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Fine-Gray models.
OS in patients who receive 6 alternated venetoclax/Daunorubincin courses of interim continuation therapy. | Up to five years for every enrolled case
  OS will be estimated using the Kaplan-Meier estimator of survival functions along with 95% confidence interval at 5 year. Standard error will be estimated using the default procedure in R. Follow up of the historical comparison cohort (CCCG-ALL-2020 and 2015) will continue during the course of the current trial. Comparisons of OS will be performed using two-sided log-rank test. Multivariable regression modeling including trial (CCCGALL-2025 vs. 2020 or 2015) and other known prognostic factors as main effects may also be performed, using the Cox models.
To compare grade 3 or higher adverse effects (AEs; CTCAE v5.0) and estimate their cumulative incidences | Up to 30 days after last dose of study treatment
  Proportions of grade-3 or higher AEs in each treatment phase will be estimated by the sample proportions along with exact 95% confidence intervals. Cumulative incidences of various grade-3 or higher AEs throughout therapy will be estimated by the Kalbafleisch-Prentice method; death, relapse and other events rendering off therapy before completion are regarded as competing risks.

OTHER OUTCOMES:
measurable residual diseases (MRD) positivity by next-generation sequencing of immunoglobulin gene(IgH NGS) after blinatumomab-HDMTX therapy between the two randomized arms [2*(14-day blinatumomab + HDMTX*2)] and [28-day blinatumomab + HDMTX*4]. | Up to five years
  Proportions of patients with positive IgH NGS MRD in each arm will be estimated by the sample proportion along with the 95% confidence interval. The NGS MRD positive proportions will be compared by the two-sample z test. If the NGS MRD positive proportions are very low in one or both arms, Fisher's exact test will be applied.
Cellular immune-status prior to Blinatumomab-HDMTX consolidation therapy | At the end of induction
  Descriptive statistics on T lymphocytes functions (exhaustion, activation, TCR diversity, etc.) including correlation coefficients (Pearson's or Spearman's) and regression modeling including possibly longitudinal data models will be applied as appropriate to analyze the biological associations.
Cellular immune functions after blinatumomab-HDMTX consolidation | Up to 2 years
  Descriptive statistics on T lymphocytes functions (exhaustion, activation, TCR diversity, etc.).including correlation coefficients (Pearson's or Spearman's) and regression modeling including possibly longitudinal data models will be applied as appropriate to analyze the biological associations.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC
Locations (26):
- China (25):
  - Anhui Medical University Second Affiliated Hospital, Hefei, Anhui
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Children's Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Xi'an Northwest Women and Children Hospital, Xi’an, Shanxi
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC, Tianjin, Tianjin Municipality
  - Chongqing Medical University Affiliated Children's Hospital, Chongqing
  - Children's Hospital of Fudan University, Shanghai
  - Shanghai Children's Hospital, Shanghai
  - Shanghai Children's Medical Cener, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shenzhen Children's Hospital, Shenzhen
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
1. Demographic Data: Age, sex, and other relevant baseline characteristics.
  2. Treatment Information: Data on interventions received by participants, including dosage, treatment cycles, and duration.
  3. Outcome Measures: Detailed information on primary and secondary outcome measures, such as response rates, survival rates, adverse events, and any the pre-specified endpoints.
  4. Adverse Events: Data on all reported adverse events, including severity, duration, and outcome.
  5. Laboratory Data: Results from laboratory tests, such as blood counts, biochemical markers, or molecular analysis.
  6. Medical History: Pre-existing conditions, comorbidities, and prior treatments or interventions.
  7. Vital Signs: relevant physiological data.
  8. Efficacy and Safety Data: Any data relating to the efficacy (e.g., event-free survival) and safety (e.g., adverse effects) of the treatment.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available upon publication of the primary trial results or after trial completion, whichever occurs first, starting on 2030, and will remain accessible for 5 years.
Access Criteria: Researchers, healthcare professionals who meet the criteria for access (e.g., academic researchers conducting secondary analyses or regulatory bodies reviewing safety data) will be able to request access to de-identified IPD and supporting information. Access will be facilitated through clinical trials.gov/emailing to PI, where users can submit a request and provide a research proposal. Data access will be granted after a formal review and approval process, subject to compliance with the data-sharing agreement and confidentiality terms.
URL: http://cccg.nipher.com/cccg/

REFERENCES:
- [Background] Middelmann HU, Sorba L, Hinkel V V, Horn K. Valence-band structure of alpha -Sn determined by angle-resolved photoemission. Phys Rev B Condens Matter. 1987 Jan 15;35(2):718-722. doi: 10.1103/physrevb.35.718. No abstract available. PMID 9941458
- [Background] Toft N, Birgens H, Abrahamsson J, Griskevicius L, Hallbook H, Heyman M, Klausen TW, Jonsson OG, Palk K, Pruunsild K, Quist-Paulsen P, Vaitkeviciene G, Vettenranta K, Asberg A, Frandsen TL, Marquart HV, Madsen HO, Noren-Nystrom U, Schmiegelow K. Results of NOPHO ALL2008 treatment for patients aged 1-45 years with acute lymphoblastic leukemia. Leukemia. 2018 Mar;32(3):606-615. doi: 10.1038/leu.2017.265. Epub 2017 Aug 18. PMID 28819280
- [Background] Teachey DT, Pui CH. Comparative features and outcomes between paediatric T-cell and B-cell acute lymphoblastic leukaemia. Lancet Oncol. 2019 Mar;20(3):e142-e154. doi: 10.1016/S1470-2045(19)30031-2. PMID 30842058
- [Background] Pui CH, Yang JJ, Hunger SP, Pieters R, Schrappe M, Biondi A, Vora A, Baruchel A, Silverman LB, Schmiegelow K, Escherich G, Horibe K, Benoit YC, Izraeli S, Yeoh AE, Liang DC, Downing JR, Evans WE, Relling MV, Mullighan CG. Childhood Acute Lymphoblastic Leukemia: Progress Through Collaboration. J Clin Oncol. 2015 Sep 20;33(27):2938-48. doi: 10.1200/JCO.2014.59.1636. Epub 2015 Aug 24. PMID 26304874
- [Background] Pieters R, de Groot-Kruseman H, Van der Velden V, Fiocco M, van den Berg H, de Bont E, Egeler RM, Hoogerbrugge P, Kaspers G, Van der Schoot E, De Haas V, Van Dongen J. Successful Therapy Reduction and Intensification for Childhood Acute Lymphoblastic Leukemia Based on Minimal Residual Disease Monitoring: Study ALL10 From the Dutch Childhood Oncology Group. J Clin Oncol. 2016 Aug 1;34(22):2591-601. doi: 10.1200/JCO.2015.64.6364. Epub 2016 Jun 6. PMID 27269950
- [Background] Moricke A, Zimmermann M, Valsecchi MG, Stanulla M, Biondi A, Mann G, Locatelli F, Cazzaniga G, Niggli F, Arico M, Bartram CR, Attarbaschi A, Silvestri D, Beier R, Basso G, Ratei R, Kulozik AE, Lo Nigro L, Kremens B, Greiner J, Parasole R, Harbott J, Caruso R, von Stackelberg A, Barisone E, Rossig C, Conter V, Schrappe M. Dexamethasone vs prednisone in induction treatment of pediatric ALL: results of the randomized trial AIEOP-BFM ALL 2000. Blood. 2016 Apr 28;127(17):2101-12. doi: 10.1182/blood-2015-09-670729. Epub 2016 Feb 17. PMID 26888258
- [Background] Leung KT, Cai J, Liu Y, Chan KYY, Shao J, Yang H, Hu Q, Xue Y, Wu X, Guo X, Zhai X, Wang N, Li X, Tian X, Li Z, Xue N, Guo Y, Wang L, Zou Y, Xiao P, He Y, Jin R, Tang J, Yang JJ, Shen S, Pui CH, Li CK. Prognostic implications of CD9 in childhood acute lymphoblastic leukemia: insights from a nationwide multicenter study in China. Leukemia. 2024 Feb;38(2):250-257. doi: 10.1038/s41375-023-02089-3. Epub 2023 Nov 25. PMID 38001171
- [Background] Jeha S, Pei D, Choi J, Cheng C, Sandlund JT, Coustan-Smith E, Campana D, Inaba H, Rubnitz JE, Ribeiro RC, Gruber TA, Raimondi SC, Khan RB, Yang JJ, Mullighan CG, Downing JR, Evans WE, Relling MV, Pui CH. Improved CNS Control of Childhood Acute Lymphoblastic Leukemia Without Cranial Irradiation: St Jude Total Therapy Study 16. J Clin Oncol. 2019 Dec 10;37(35):3377-3391. doi: 10.1200/JCO.19.01692. Epub 2019 Oct 28. PMID 31657981
- [Background] Hunger SP, Lu X, Devidas M, Camitta BM, Gaynon PS, Winick NJ, Reaman GH, Carroll WL. Improved survival for children and adolescents with acute lymphoblastic leukemia between 1990 and 2005: a report from the children's oncology group. J Clin Oncol. 2012 May 10;30(14):1663-9. doi: 10.1200/JCO.2011.37.8018. Epub 2012 Mar 12. PMID 22412151
- [Background] Escherich G, Zimmermann M, Janka-Schaub G; CoALL study group. Doxorubicin or daunorubicin given upfront in a therapeutic window are equally effective in children with newly diagnosed acute lymphoblastic leukemia. A randomized comparison in trial CoALL 07-03. Pediatr Blood Cancer. 2013 Feb;60(2):254-7. doi: 10.1002/pbc.24273. Epub 2012 Sep 4. PMID 22948968
- See also: data collecting website — http://cccg.nipher.com/cccg/
- Available data/document: Individual Participant Data Set: CCCG-ALL — http://cccg.nipher.com/cccg/ — CCCG-ALL-2025 DATASET